CLINICAL TRIAL: NCT03003871
Title: A Randomized Clinical Trial on the Effect of Powered Toothbrushing and an Antimicrobial Mouth Rinse on Dental Plaque, Pathogenic Microorganisms and Health of Stroke Survivors During Rehabilitation.
Brief Title: Oral Health Promotion Interventions Amongst Stroke Survivors During Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Tung Wah Hospital (Other)
Responsible Party: Principal Investigator, Professor Colman Patrick McGrath, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GRF774012
Record Dates: First submitted 2016-09-09; First posted 2016-12-28 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Stroke
Keywords: stroke; randomized controled clinical trial; oral health promotion
MeSH Terms: conditions — Stroke | interventions — Toothpastes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- advanced oral hygiene care programmes (Experimental): participants were provided with a powered toothbrush (Oral-B® AdvancePowerTM 400 series), 0.2% chlorhexidine gluconate mouth rinse, 10 mls twice daily (CorsodylPTMP), standardized toothpaste (Colgate Maximum Cavity Protection) and oral hygiene instruction.
  Interventions: Device: Powered toothbrush; Other: Toothpaste; Other: 0.2% chlorhexidine gluconate mouth rinse
- conventional oral hygiene care programme (Active Comparator): participants were provided with a manual toothbrush (Oral-B® Pro-Health All-In-One), supply of a standardized toothpaste (Colgate Maximum Cavity Protection®) and oral hygiene instruction
  Interventions: Device: Manual toothbrush; Other: Toothpaste

INTERVENTIONS:
Device: Powered toothbrush — Oral-B® AdvancePowerTM 400 series
  Arms: advanced oral hygiene care programmes
Device: Manual toothbrush — Oral-B® Pro-Health All-In-One
  Arms: conventional oral hygiene care programme
Other: Toothpaste — Colgate Maximum Cavity Protection®
Other: 0.2% chlorhexidine gluconate mouth rinse — CorsodylPTMP
  Arms: advanced oral hygiene care programmes

SUMMARY:
Stroke is the second most common cause of death worldwide and is the predominant cause of permanent disability among older people. The mouth becomes a very unhealthy place after stroke, where yeasts and pathogenic bacteria multiply at an accelerated rate. Poor oral hygiene results in increased dental plaque, gingival bleeding, and the harbouring of oral opportunistic pathogens. Dental plaque acts as a reservoir of pathogenic microorganisms which results in additional oral health problems and also can cause life-threatening medical complications; most notably aspiration pneumonia and/or recurrent stroke. The first six months following stroke is a particular vulnerable period to survive.

Removal of dental plaque and its associated pathogenic microorganisms is challenging in this compromised state of reduced manual dexterity and weak state following a stroke. Powered (electric) toothbrushes can be of assistance in plaque removal in frail elders. For more resistant oral pathogens, anti-plaque/anti-microbial mouthrinses can offer additional help in controlling dental plaque and thereby prevent harbouring potentially life threatening oral pathogens. Over the years the Faculty of Dentistry and the Stroke Rehabilitation Unit of the Department of Medicine in Hong Kong have been actively working together to address the problems of oral health associated with stroke; and specifically the challenge of safeguarding the life and health of stroke survivors during the vulnerable rehabilitation period. We are now proposing to involve stroke patients during out-patient rehabilitation in a randomized clinical trial to test the effectiveness of powered tooth brushing and a chlorhexidine anti-microbial mouthrinse in reducing dental plaque accumulation and oral pathogens; and how this affects their general and oral health status. We anticipate that all participants will benefit from the oral health promotion initiatives and that the advantages will be long lasting. We expect to demonstrate a 'gold standard' of oral health preventive care, as part of stroke rehabilitation, that can reduce (or has potential to reduce) serious medical complications after a stroke. If proven effective this oral health preventive care regime (which is relatively easy to implement and at low cost) could widely be adopted in stroke rehabilitation globally.

DETAILED DESCRIPTION:
The study population in this clinical trial will be patients with moderate to severe stroke undergoing further stroke rehabilitation by returning regularly to the Day Rehabilitation Center (on an out-patient basis) of the Rehabilitation Unit at Tung Wah Hospital (TWH). The TWH Rehabilitation Unit, Sheung Wan, Hong Kong has been selected as the study site because it serves a major urban area in Hong Kong. TWH is a medical teaching hospital, patient medical care is standardized and a comprehensive set of records is compiled during stroke rehabilitation. Around 500 patients with acute stroke are admitted annually to the Rehabilitation Unit. The majority of the patients are stabilized (for up to 7 days) at Queen Mary Hospital, a major teaching hospital for treating acute medical conditions, prior to admission to the Rehabilitation Unit. On admission to the Rehabilitation Unit, each stroke patient undergoes a comprehensive medical assessment that includes a functional disability assessment using the modified Barthel Index and a rehabilitation programme is formulated. Following hospital discharge, patients requiring further rehabilitation return regularly to the Day Rehabilitation Center on an out-patient basis. Stroke patients deemed fit for discharge from the Rehabilitation Unit will be invited to participate in the study in accordance with the inclusion & exclusion criteria.

The key outcome variable of this clinical trial is the dental plaque level (the key reservoir for oral pathogens). In a previous observational study we conducted among stroke survivors, the mean PI score was 2.1 (standard deviation [SD]=0.51) at discharge and 1.9 (SD=0.56) at 6 months, yielding a change score of 0.21 (SD=0.46). On the basis of this study, and proposing a difference in plaque change scores of at least 0.3 between baseline to follow-up (and also between groups) and with the standard deviation set at 0.46, then the number of study subjects that would be required is 38 per group, based on 80% power and the statistical significance level set at 0.05. Anticipating a 20% dropout rate over the course of the clinical trial, the initial sample size for each treatment group is proposed as 47 patients per group (94 subjects in total).

Assessments of clinical oral health status, presence of oral opportunistic pathogens and subjective oral health were conducted at baseline, 3 month and 6 month. All assessments were performed in the TWH Day Rehabilitation Center. Compliance was also assessed. Data will be stored on a computer (and backed up on a compact disc) in the Faculty of Dentistry, The University of Hong Kong. Professor Colman McGrath (Principle Investigator) will be responsible for its safekeeping. All data will be kept until analyses have been performed and all research manuscripts have been accepted for publication. The data will then be destroyed.

The statistics software packages SPSS 21 for Windows (SPSS Inc., Chicago, USA) and STATA 13.0 for Windows (IBM) were used in all statistical tests. Both per-protocol (PP) and intention-to-treat (ITT) analyses was employed for both primary and secondary outcomes. In bivariate analyses, within and between groups comparisons were made over the clinical trial period. When the outcome variables were continuous and followed a normal distribution, paired t test for related samples were performed to determine significant differences over time. Student t-test for independent samples was performed to compare the mean of the outcomes between intervention groups at baseline and follow-up review. When the outcome variables were continuous but did not follow a normal distribution as detected by normality test, Wilcoxon Signed Rank test (a non-parametric equivalence of the paired t test for related samples) was performed to determine significant differences over time. Mann Whitney U test (a non-parametric equivalence of the t test for independent samples) was employed to compare difference in the rank of outcomes between intervention groups at baseline and follow-up. When the outcome variables were categorical, McNemar test were performed to identify changes in prevalence over time and Chi-square test was employed to compare variations in prevalence between intervention groups at baseline and follow up.

Regression analyses were employed to address the effect of potential explanatory factors for outcomes. When conducting the regression analysis, method of Last Observation Carried Forward (LOCF) was employed to deal with missing outcomes at follow-up reviews. Linear regression was adopted when the dependent variables were continuous and residuals of the regression followed a normal distribution. Negative binomial regression was adopted when the continuous dependent variables had over-dispersed count data. Logistic regression was adopted when the dependent variables were binary. Since the effect of intervention on the outcomes was of our core interest, the model fitting adopted a forward-wald method with the factor of intervention fixed in the model and one of the other explanatory factors added into the model each time. Each time the coefficient of the independent variables with the smallest significant p value (significance level p<0.05) was entered into the regression model. The model fitting process was repeated again until no more independent variable had significant p values.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to participate in the Day Rehabilitation Center rehabilitation programme;
2. Had moderate to severe functional disability- Barthel Index (BI) scores of <70;
3. Able to follow a one-step command (as an assessment of communication)

Exclusion Criteria:

1. edentulous;
2. more than mild cognitive ability- Mini Mental State Examination (MMSE) less than18;
3. had an indwelling naso-gastric feeding tubes.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
plaque index (PI) at 3 months | 3 months
  The PI was charted on all permanent teeth and assessed at six sites per tooth at 3 months. The criteria for the Silness and Löe Plaque are as following: 0 = No plaque detected with probe; 1 = Plaque not visible by unaided eye but detectable with probe; 2 = Moderate amount of plaque. Plaque visible to unaided eye; 3 = Abundance of plaque. The percentage of tooth sites with moderate to abundant plaque (PI score: 2 or 3) was calculated for each subject.

SECONDARY OUTCOMES:
prevalence and viable counts of oral opportunistic pathogens at 3 months | 3 months
  The oral rinse samples were collected at 3 months. The oral rinse technique was used to detect oral opportunistic pathogens colonization in the whole oral cavity. A spiral plater (Spiral Systems Marketing Limited, Maryland, USA) was employed to inoculate the samples onto four selective cultural medium. Isolates on the above selective cultural medium were presumptively identified by colony morphology and the Gram stain method, and quantified by colony forming units (cfu/ml).
prevalence and viable counts of oral opportunistic pathogens at 6 months | 6 months
  The oral rinse samples were collected at 6 months. The oral rinse technique was used to detect oral opportunistic pathogens colonization in the whole oral cavity. A spiral plater (Spiral Systems Marketing Limited, Maryland, USA) was employed to inoculate the samples onto four selective cultural medium. Isolates on the above selective cultural medium were presumptively identified by colony morphology and the Gram stain method, and quantified by colony forming units (cfu/ml).
health-related quality of life (HRQL) at 3 months | 3 months
  The subjective health assessment included generic health-related quality of life (HRQL) and oral health-related quality of life (OHRQL) assessments. This consisted of the Cantonese versions of the Short Form Health Survey 12 (SF-12), the Oral Health Impact Profile 14 (OHIP-14), the Geriatric Oral Health Assessment Index (GOHAI).
health-related quality of life (HRQL) at 6 months | 6 months
  The subjective health assessment included generic health-related quality of life (HRQL) and oral health-related quality of life (OHRQL) assessments. This consisted of the Cantonese versions of the Short Form Health Survey 12 (SF-12), the Oral Health Impact Profile 14 (OHIP-14), the Geriatric Oral Health Assessment Index (GOHAI).
plaque index (PI) at 6 months | 6 months
  The PI was charted on all permanent teeth and assessed at six sites per tooth at 6 months. The criteria for the Silness and Löe Plaque are as following: 0 = No plaque detected with probe; 1 = Plaque not visible by unaided eye but detectable with probe; 2 = Moderate amount of plaque. Plaque visible to unaided eye; 3 = Abundance of plaque. The percentage of tooth sites with moderate to abundant plaque (PI score: 2 or 3) was calculated for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Colman McGrath, PhD, Principal Investigator — Facluty of Dentistry, the University of Hong Kong

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Lam CL, Tse EY, Gandek B. Is the standard SF-12 health survey valid and equivalent for a Chinese population? Qual Life Res. 2005 Mar;14(2):539-47. doi: 10.1007/s11136-004-0704-3. PMID 15892443
- [Background] Wong MC, Liu JK, Lo EC. Translation and validation of the Chinese version of GOHAI. J Public Health Dent. 2002 Spring;62(2):78-83. doi: 10.1111/j.1752-7325.2002.tb03426.x. PMID 11989210
- [Background] Wong MC, Lo EC, McMillan AS. Validation of a Chinese version of the Oral Health Impact Profile (OHIP). Community Dent Oral Epidemiol. 2002 Dec;30(6):423-30. doi: 10.1034/j.1600-0528.2002.00013.x. PMID 12453113
- [Background] Zhu HW, McMillan AS, McGrath C, Li LS, Samaranayake LP. Oral carriage of yeasts and coliforms in stroke sufferers: a prospective longitudinal study. Oral Dis. 2008 Jan;14(1):60-6. doi: 10.1111/j.1601-0825.2006.01347.x. PMID 18173450